CLINICAL TRIAL: NCT01642875
Title: Early Oral Versus Enteral Nutrition After Pancreatoduodenectomy for Periampullary Tumors: a Prospective, Randomized, Controlled Clinical Trial
Brief Title: Early Oral Versus Enteral Nutrition After Pancreatoduodenectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PerOsEnteral1
Record Dates: First submitted 2012-07-09; First posted 2012-07-17 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Pancreatic Cancer; Cancer of the Duodenum; Cholangiocarcinoma; Chronic Pancreatitis
Keywords: Periampullary tumor; Chronic pancreatitis; Pancreatoduodenectomy; Oral Nutrition; Enteral Nutrition
MeSH Terms: conditions — Pancreatic Neoplasms; Duodenal Neoplasms; Cholangiocarcinoma; Pancreatitis, Chronic | interventions — Enteral Nutrition; Nutritional Status; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EN (Experimental): early enteral nutrition with standard enteral formulas administered through a nasojejunal tube
  Interventions: Other: Enteral nutrition
- PerOs (Active Comparator): early oral nutrition with hospital diets and oral formulas
  Interventions: Other: Oral nutrition

INTERVENTIONS:
Other: Enteral nutrition — Standard enteral diet is administered through a nasojejunal tube. Enteral nutrition is started on the 1st postoperative day and increased daily by 20-40 ml up to the estimated level.
  Other Names: standard enteral formula
  Arms: EN
Other: Oral nutrition — Oral diet is started from the 2nd postoperative day and oral intake is advanced as tolerated
  Other Names: oral diet
  Arms: PerOs

SUMMARY:
Pancreatoduodenectomy carries high morbidity rates even in high-volume centers. Postoperative complications often preclude or delay adequate oral nutrition and nutritional support may be required. However, the role of perioperative nutritional supplementation in well-nourished patients remains controversial.

The purpose of this study is to compare the influence of early enteral and oral nutrition on postoperative course and complications after pancreatoduodenectomy.

96 patients undergoing pancreatoduodenectomy will be randomized to receive early enteral nutrition (EN group) or early oral nutrition (PerOs group). The EN group will receive standard enteral diet administered through a nasojejunal tube. Enteral nutrition will be started on the 1st postoperative day and increased daily by 20-40 ml up to the estimated level. The PerOs group will receive oral diets beginning from the 2nd postoperative day and oral intake will be advanced as tolerated.

DETAILED DESCRIPTION:
Background & aim: Pancreatoduodenectomy carries high morbidity rates even in high-volume centers. Postoperative complications often preclude or delay adequate oral nutrition and nutritional support may be required. However, the role of perioperative nutritional supplementation in well-nourished patients remains controversial. There are not any standard protocols for nutritional support after major upper gastrointestinal surgery in these patients and postoperative nutritional regimens depend mainly upon surgeon's or center preference.

Patients undergoing pancreatoduodenectomy often begin oral intake a week after operation and enteral or parenteral nutrition is used to cover the daily caloric requirements during this period, although their role still remains questionable. The safety of early oral nutrition has been confirmed in the majority of gastrointestinal procedures. However, pancreatic surgeons are quite reluctant to advance oral diet within the first postoperative week after pancreatoduodenectomy due to fear of anastomosis breakdown or delayed gastric emptying syndrome. These two postoperative nutritional regimens, early oral vs. early enteral nutrition, have not been sufficiently evaluated in a prospective, randomized study.

Material and Methods: 96 patients undergoing pancreatoduodenectomy will be randomized to receive early enteral nutrition (EN group) or early oral nutrition (PerOs group). The EN group will receive standard enteral diet administered through a nasojejunal tube. The enteral nutrition will be started on the 1st postoperative day and increased daily by 20-40 ml up to the estimated level. The PerOs group will receive oral diets beginning from the 2nd postoperative day and oral intake will be advanced as tolerated.

Purpose: The purpose of this study is to compare the influence of early enteral and oral nutrition on postoperative course and complications after pancreatoduodenectomy.

ELIGIBILITY:
Inclusion Criteria:

* Primary periampullary tumor
* R0, R1 resection
* Chronic pancreatitis requiring pancreatoduodenectomy

Exclusion Criteria:

* Metastatic tumor
* Locally unresectable tumor
* Previous gastric resection
* ASA IV-V
* Age under 18 years
* Preoperative complete parenteral or enteral feeding
* Immunosuppressive therapy before operation
* Severe malnutrition
* Lack of the patient's consent for the trial participation, feeding tube insertion or epidural analgesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of delayed gastric emptying | 30 days after operation

SECONDARY OUTCOMES:
Overall morbidity rate | 60 days after operation
Perioperative mortality rate | 60 days after operation
Postoperative hospital stay length | 60 days after operation
Time to full oral nutrition | 60 days after operation
Time to resolution of paralytic ileus | 7 days after operation
Rehospitalization rate | 30 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Słodkowski, MD, Study Director — Medical University of Warsaw; Marek Wronski, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Sp Csk Wum, Warsaw, Poland